CLINICAL TRIAL: NCT00677456
Title: Postoperative Life Quality Evaluation of Four Reconstructions After Total Gastrectomy
Brief Title: Evaluation of Four Reconstructions After Total Gastrectomy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Collaborators: Air Force Military Medical University, China (Other)
Responsible Party: He XianLi/director of department of Gastrointestinal Surgery, Tang-Du Hospital, Department of Gastrointestinal Surgery, Tang-Du Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TDH00431
Record Dates: First submitted 2008-05-12; First posted 2008-05-14 (Estimated); Last update posted 2008-05-14 (Estimated); Status verified 2008-01

CONDITIONS: Gastric Cancer; Nutrition
Keywords: Gastric Cancer; total gastrectomy; reconstruction; life quality
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): Patients will receive R-Y reconstruction after total gastrectomy as intervention
  Interventions: Procedure: R-Y reconstruction after total gastrectomy
- 2 (Active Comparator): Patients will receive P-Y reconstruction after total gastrectomy as intervention
  Interventions: Procedure: P-Y reconstruction after total gastrectomy
- 3 (Active Comparator): Patients will receive Pouch reconstruction after total gastrectomy as intervention.
  Interventions: Procedure: Pouch reconstruction after total gastrectomy
- 4 (Active Comparator): Patients will receive P-I reconstruction after total gastrectomy as intervention.
  Interventions: Procedure: P-I reconstruction after total gastrectomy

INTERVENTIONS:
Procedure: R-Y reconstruction after total gastrectomy — Following curative total gastrectomy and systematic lymphadenectomy, the jejunum was divided 20 cm distal to the Treitz ligament with preservation of the nerve along the marginal vessels. The distance of the esophagojejunostomy to the jejunojejunostomy was 40 cm for the R-Y.
  Other Names: R-Y reconstruction
  Arms: 1
Procedure: P-Y reconstruction after total gastrectomy — Following curative total gastrectomy and systematic lymphadenectomy, the jejunum was divided 20 cm distal to the Treitz ligament with preservation of the nerve along the marginal vessels. The distance of the esophagojejunostomy to the jejunojejunostomy was 40 cm for the P-Y.
  Other Names: P-Y reconstruction
  Arms: 2
Procedure: Pouch reconstruction after total gastrectomy — Following curative total gastrectomy and systematic lymphadenectomy, the jejunum was divided 20 cm distal to the Treitz ligament with preservation of the nerve along the marginal vessels. To make the jejunal pouch, jejunojejunostomy was done with a linear stapler at the antimesenteric border, the distance of the esophagojejunostomy to the jejunojejunostomy was 40 cm for the R-Y.
  Other Names: Pouch reconstruction
  Arms: 3
Procedure: P-I reconstruction after total gastrectomy — Following curative total gastrectomy and systematic lymphadenectomy, the jejunum was divided 20 cm distal to the Treitz ligament with preservation of the nerve along the marginal vessels.To make the jejunal pouch, jejunojejunostomy was done with a linear stapler at the antimesenteric border,The pouch was 20 cm long, with a 10-cm jejunal loop with the P-I.
  Other Names: P-I reconstruction
  Arms: 4

SUMMARY:
There are four capital reconstructions after total gastrectomy which is widely used in China. Life quality is the only standard to evaluate postoperative results of different reconstructions. In order to determine the best reconstruction after total gastrectomy, we designed this study to compare life qualities of four reconstructions.

ELIGIBILITY:
Inclusion Criteria:

* Patients should be younger than 80 years old with adequate renal, pulmonary, and heart functions.

Exclusion Criteria:

* death or other reason which cause information discontinue

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-02 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Patients should live for 6 months at least, and with acceptable life quality | 6 months

SECONDARY OUTCOMES:
There are significant differences among life qualities of the four reconstructions | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: XianLi He, doctor, Principal Investigator — Department of general surgery, Tangdu hospital of fourth military medical university
Locations (1):
- Department of general surgery,Tangdu hospital, Xi'an, Shaanxi, China